CLINICAL TRIAL: NCT00511849
Title: Phase I Study Of SU011248 In Combination With Paclitaxel/Carboplatin In Patients With Advanced Solid Malignancies
Brief Title: Study Of SU011248 In Combination With Paclitaxel/Carboplatin In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181050
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Carboplatin; Sunitinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: carboplatin + SU011248 (sunitinib) + paclitaxel

INTERVENTIONS:
Drug: carboplatin + SU011248 (sunitinib) + paclitaxel — AUC of 6 mg*min/mL administered as a 30-minute infusion, every 21 days for 4 cycles or until progression/unacceptable toxicity. 25 mg, 37.5 mg, or 50 mg (depending on the dose level assigned) orally taken every day or for 2 weeks and 1 week off without for 4 cycles or until progression/unacceptable toxicity. 175 mg/m2, 200 mg/m2, or 225 mg/m2 (depending on the dose level assigned), administered as a 3-hour infusion every 21 days for 4 cycles or until progression/unacceptable toxicity.
  Other Names: Paraplatin; SUTENT; Taxol

SUMMARY:
The purpose of this study is to test SU011248 (sunitinib) in combination with paclitaxel/carboplatin. This combination regimen will be tested for safety and antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of any advanced solid malignancy that is not amenable to treatment with curative intent
* Candidates for treatment with carboplatin and paclitaxel with maximum of 2 prior chemotherapy regimens
* ECOG performance status 0 or 1

Exclusion Criteria:

* Prior chemotherapy, radiation therapy or surgery within 4 weeks prior to study entry except palliative radiotherapy to non-target, metastatic lesions
* Diagnosis of any second malignancy within the past 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose (MTD) and overall safety of SU011248 when administered in combination with paclitaxel/carboplatin in patients with advanced solid tumors (ongoing) | 3 yrs

SECONDARY OUTCOMES:
Evaluate pharmacokinetic parameters of carboplatin, paclitaxel, SU011248 and its active metabolite, SU012662. Assess antitumor activity of the combination. | 3 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181050&StudyName=Study%20Of%20SU011248%20In%20Combination%20With%20Paclitaxel/Carboplatin%20In%20Patients%20With%20Advanced%20Solid%20Tumors%0A